CLINICAL TRIAL: NCT01509066
Title: Healthy Eating for Reproductive Health (HERHealth)
Acronym: HERHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014149
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Polycystic Ovarian Syndrome; Infertility; Obesity; Overweight
Keywords: vegetarian; vegan; low calorie; infertility; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Obesity; Overweight | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegan diet (Experimental): A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. We will also ask participants to keep foods low in fat and low in glycemic index.
  Interventions: Other: Diet
- Low-calorie (Active Comparator): A low-calorie diet contains all food groups. However, participants will be provided with a calorie goal which should promote weight loss.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Dietary approaches for PCOS

SUMMARY:
This study will be a 6-month intervention that is examining how different dietary approached may be useful for women with Polycystic Ovarian Syndrome (PCOS) who are attempting pregnancy, particularly by measuring changes in weight. Participants will be randomly assigned to following one of two dietary approaches for weight loss: 1) a low-calorie approach to weight loss (reducing caloric intake by approximately 500 calories per day) or 2) a low-fat, low-glycemic index vegan diet. A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. In addition, this diet will be low-glycemic index, which means you will be asked to favor foods that don't cause a quick rise in blood sugar (for example, favoring oatmeal over cornflakes for breakfast). Participants will receive counseling and supporting materials on the dietary approach you are assigned to follow. Both diets are safe and have shown to be effective ways to assist with achieving a healthy weight. The investigators hypothesize that both groups will see improvements in weight and fertility with possible greater improvements seen among participants in the vegan group.

DETAILED DESCRIPTION:
This study involves two groups. You will be randomly assigned to one of these groups (i.e. you do not have a choice for group assignment) which means your group will be assigned to you by chance, like flipping a coin. Both groups will be assigned to receive information on a dietary approach to lose weight. One group will receive instruction on a low-calorie approach to weight loss (reducing caloric intake by approximately 500 calories per day). The other group will be instructed on how to follow a low-fat, low-glycemic index vegan diet. A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. In addition, this diet will be low-glycemic index, which means you will be asked to favor foods that don't cause a quick rise in blood sugar (for example, favoring oatmeal over cornflakes for breakfast). Below are the steps in the study:

* If you are accepted into the study, you will come to the study site (USC School of Public Health) to learn more about the study and complete your consent form. If you live outside the Columbia, SC area (more than a 6o mile drive), then you may complete orientation to the study over the phone and Web. You will then be mailed a consent form which we will discuss over the phone. You can then sign the consent form (keeping one copy for yourself and having a witness sign it as well) and mail it back. Once that is received by study personnel, a copy with a research personnel's signature will be mailed back to you. You may then begin the study.
* This study will involve 3-4 in-person visits to the School of Public Health at USC's Columbia campus, each lasting less than 2 hours each.
* You will then complete some questionnaires that will measure your diet and physical activity levels at home from a computer.
* You will come back for a meeting to have your weight, height, waist, and hip circumference measured. You will then be randomly assigned to one of the two groups: calorie controlled group or vegan diet group. You will receive a one-hour overview of the diet you have been assigned to and be provided with materials on this diet.
* During the study, we will ask you to complete a weekly questionnaire which will assess if you are following the diet, your weight, and ask for information on your menstrual cycle. This will take approximately 5 minutes to complete.
* You will then be provided individualized feedback each week via e-mail on your progress, along with a weekly lesson on the topic for the week.
* You will also have access to a group website (a private Facebook group) that will provide group support. Participation using this group is optional.
* You will be provided with test strips to monitor ovulation each month and pregnancy tests (1 per month) to monitor pregnancy status. You will report these results to us via online survey.
* Study personnel will host a weekly 30 minute webinar for your diet group online. This will take place after work time on a weekday. Make-up sessions by phone during the work day will be available.
* At 3 months, you will be asked to complete another set of questionnaires from home and return to our study site for your weight, waist, and hip circumference measurements. You will receive a $10 incentive for completing the 3-month assessment. You will also receive a $5 incentive each month that you provide your menstrual cycle data (using the test strips) and pregnancy tests results-which you will receive at the 3 month meeting (for a total of $25 possible at month 3).
* You will then continue the study for the next 3 months.
* At study completion (6 months), you will complete the last set of questionnaire (online from home). Also, you will come to a follow-up assessment to be weighed, have your waist and hip circumference measured, and to receive your incentive for participating ($10 +$5/month of each menstrual cycle data submitted for a total of $25 possible).
* If you become pregnant during the course of the study, you will be advised to consult your care provider. Because this is a weight loss study, we cannot allow continued participation but would like to record your weight measurement and other questionnaire data prior to study discontinuation. If you choose to continue to follow your assigned dietary approach, we can provide information on the diet to your physician, who can advise you on how to proceed.
* Participants in both groups will be asked to take a daily prenatal vitamin (or other reliable source of vitamin B-12) over the course of the study.
* During the study, we will ask you to keep your physical activity levels constant (keep your levels the same as what you were doing at study entry).

ELIGIBILITY:
Inclusion Criteria:

* Women must meet the following criteria:

  * have been attempting pregnancy for at least 6 months
  * is not currently pregnant
  * has a clinical diagnosis of PCOS
  * is not on oral medications for insulin resistance (such as metformin) or, if currently on such a medication, has been on the medication at a stable dose for at least 3 months
  * willing not use fertility-enhancing medications over the 6-month study (with the exception of oral medications, such as clomiphene citrate, as directed by their physician)
  * willing to be randomized to either dietary condition and able to make weekly meetings.

Exclusion Criteria:

Participants should not be in this study if they meet any of the following criteria:

* have not been diagnoses with polycystic ovarian syndrome
* have been trying to conceive less than 6 months
* have a Body Mass Index less than 25 or greater than 45 kg/m2
* are currently pregnant
* are younger than 18 or older than 35 years of age
* are a smoker
* are unable to come to the Columbia, SC area at least 3-4 times in a 6 month time period for assessments
* don't have access to the Internet and a computer
* don't have access to a scale for self-monitoring weight
* aren't willing to be randomized to either group
* have a psychiatric disease, drug or alcohol dependency, or uncontrolled thyroid condition
* have a major health condition, such as heart conditions, diabetes, and past incidence of stroke
* unable to receive consent from your doctor to participate if you currently are on blood pressure medications, have issues with dizziness, or have bone or joint issues
* have an eating disorder
* currently participating in a weight loss program or taking weight loss medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Body weight changes | 6 months
  body weight will be assessed at 0, 3, and 6 months

SECONDARY OUTCOMES:
Pregnancy rates | 6 months
  We will measure any occurrences of pregnancy over the course of the study
Menstrual cycle length | 6 months
  We will measure changes in the length of menstrual cycles over the course of the 6 month study

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, MS, RD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States